CLINICAL TRIAL: NCT01590303
Title: A Pilot Study Examining the Efficacy of Vitamin C Administration in Septic Patients.
Brief Title: Outcome Following Vitamin C Administration in Sepsis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Sharpe, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UWO HSREB #18803
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Severe Sepsis
Keywords: severe sepsis
MeSH Terms: conditions — Sepsis | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C (Experimental): Intravenous Vitamin C will be administered (1 gram) every 8 hours for 28 days or discharge from intensive care unit
  Interventions: Drug: Vitamin C
- placebo (Placebo Comparator): placebo vehicle administered in same fashion as active treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin C — Intravenous Vitamin C 1 gram every 8 hours for 28 days or discharge from intensive care unit
  Arms: Vitamin C
Drug: placebo — placebo vehicle administered to match volume of treatment drug every 8 hours for 28 days or until discharge from ICU
  Arms: placebo

SUMMARY:
This study is designed to determine if Vitamin C administration to septic patients will result in an improvement in organ dysfunction which occurs during a septic illness.

Hypothesis: 1. Vitamin C in sepsis will reduce the injury to organs 2. Vitamin C will reduce the length of time on a ventilator, length of stay in the intensive care unit and in hospital.

DETAILED DESCRIPTION:
This study will measure biomarkers of inflammation, coagulation and oxidative stress. These biomarkers have been shown to be increased during periods of oxidative stress eg post-operative, trauma, sepsis. The investigators will determine if Vitamin C administration decreases oxidative stress and as a result, a decrease in the markers of organ dysfunction eg SOFA Scores. Ultimately, if the investigators show a decrease in injury to organs, will this result in a better outcome for patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe sepsis
* admitted to the intensive care unit

Exclusion Criteria:

* allergy to Vitamin C
* history of kidney stones
* glucose-6-phosphate dehydrogenase deficiency
* history of iron overload/hemochromatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Sequential organ function assessment score (SOFA) | 28 days or discharge from intensive care unit
  Scoring system to determine the extent of a patient's organ function or rate of failure. The score based on 6 different scores; one each for respiratory, hepatic, cardiovascular, renal, coagulation, neurologic.

SECONDARY OUTCOMES:
Biomarkers as a measure of coagulation, inflammation and oxidative stress. | 28 days or discharge from intensive care unit
  Vitamin C Assays - Plasma/WBC Cytokines (8- plex) Adhesion Molecules Procalcitonin C-Reactive Protein,H igh Sensitivity High Density Lipoprotein Cholesterol Tbars F2 isoprostane Neutrophil elastase Thrombomodulin Free DNA HIF-1α

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Sharpe, MD FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada